CLINICAL TRIAL: NCT06537895
Title: Eating Disorders Clinical Research Network
Acronym: EDCRN
Status: Not yet recruiting | Type: Observational
Sponsor: King's College London (Other)
Collaborators: South London and Maudsley NHS Foundation Trust (Other); Imperial College London (Other); University College, London (Other); Oxford Health NHS Foundation Trust (Other Government); NHS Greater Glasgow and Clyde (Other); Birmingham Women's and Children's NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: RE22072; MR/X030539/1 (Other Grant/Funding Number: Medical Research Council); 341570 (Other: Health Research Authority)
Record Dates: First submitted 2024-07-23; First posted 2024-08-05 (Actual); Last update posted 2024-08-05 (Actual); Status verified 2024-07

CONDITIONS: Eating Disorders
MeSH Terms: conditions — Feeding and Eating Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: EDCRN questionnaires — Participants will complete questionnaires and have blood and other physical tests as specified in the EDCRN dataset.

SUMMARY:
UK Eating Disorder services are facing unprecedented demand, with effective service delivery hampered by inadequate resources, fragmented services and variable care pathways. Individuals with eating disorders, families and clinicians all agree on the critical need to improve care pathways and treatment, leading to better outcomes.

Eating disorders are serious, complex conditions influenced by a blend of biological, psychological, and environmental factors. The approach of this project is grounded in the "biopsychosocial" model. Recently, anorexia research confirms a genetic component, with biological, metabolic, and psychological mechanisms at play. Further biological research across eating disorders could allow a better understanding of the mechanisms underlying eating disorder development and better, more personalised treatments.

This project will test the feasibility of establishing a UK-wide NHS research network spanning child and adult eating disorder services to enable a step change in the ability to conduct eating disorder research. It will help address fragmentation and facilitate novel biological, psychological, and social research collaborations. The data the investigators gather will be open to all researchers for data analyses, and the collaborations established will form a collaborative network to enable future clinical trials, experimental medicine and psychology.

The study will be conducted at child and adult eating disorder services who opt to join the Network. Participants will be patients receiving treatment for an eating disorder at one of the participating services, and their parents/guardians if applicable.

Participants will complete questionnaires and have blood and other physical tests as specified in the EDCRN dataset. The study will last until 29th October 2026 (the end of the current funding period) and/or when a participant is discharged from treatment, whichever is sooner. For participants discharged before the study ends, there will be an opportunity for patients to complete optional follow-up questionnaires on a periodic basis.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have been diagnosed with an eating disorder under at least 1 of the criteria specified in the DSM-5 and/or ICD-9, 10 or 11.
* Patients who are receiving treatment as inpatients, day-patients or outpatients at a CAMHS or Adult service who is participating in the EDCRN.
* Patients who are receiving treatment in the UK.

OR:

* Parents/guardians of patients who have been diagnosed with an eating disorder under at least 1 of the criteria specified in the DSM-5 and/or ICD-9, 10 or 11.
* Parents/guardians of patients who are receiving treatment as inpatients, day-patients or outpatients at a CAMHS or Adult service who is participating in the EDCRN.
* Parents/guardians of patients who are receiving treatment in the UK.

Exclusion Criteria:

* Individuals who do not meet the criteria specified above will be considered ineligible to participate in the EDCRN.

Ages: 8 Years to 100 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: The study population are individuals who are receiving treatment for an eating disorder(s) at a UK-based eating disorder service which is part of the EDCRN and (if desired by the patient and caregiver) their parents/guardians.
Sampling Method: Non-Probability Sample
Enrollment: 12000 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2026-10-29 (Estimated); Study Completion 2026-10-29 (Estimated)

PRIMARY OUTCOMES:
EDCRN dataset | 29th October 2026
  The existence of a well-described dataset (maintained by at >50% eating disorder services across the UK) of eating disorder presentation, treatment, outcomes, demographics, social risk factors, and blood test results which can be accessed (with appropriate permissions) by researchers and others for the purposes of addressing novel research questions and facilitating service improvement efforts.
  The EDCRN dataset comprises the following parameters:
  * ED Behaviours/cognitions
  * Depression
  * Anxiety
  * Autism
  * OCD
  * Perfectionism
  * Emotional regulation
  * Psychosocial impairment
  * Adverse experiences
  * Self-injurious behaviour
  * Food insecurity
  * Physical/somatic symptoms
  * ADHD
  * Alcohol use
  * PTSD symptoms
  * Self-administered comorbidity
  * Weight stigma
  * Treatment experience
  * Comorbidities
  * Caregiver impact
  * Weight history
  * Muscle power
  * Endocrine function
  * Liver function
  * Cardiac function
  * Electrolytes
  * Bone health
  * Demographics

SECONDARY OUTCOMES:
Data on treatment effects | 29th October 2026
  Data which provides insights into treatment moderators and mediators for different demographic groups.
Genetic Biomarkers | 29th October 2026
  Indicators of genetic biomarkers of treatment response.
Socio-economic influences | 29th October 2026
  Data which indicates socio-economic factors (e.g. the local food environment) influencing ED development, maintenance and outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Gerome Breen, PhD, Principal Investigator — King's College London (KCL); Karina Allen, PhD, Principal Investigator — South London and Maudsley NHS Foundation Trust (SLaM)